CLINICAL TRIAL: NCT03562611
Title: Flurbiprofen Axetil and Nalbuphine for Postoperative Pain and Discomfort After Orbital Decompression
Brief Title: Postoperative Pain and Discomfort After Orbital Decompression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huijing Ye, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201806
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Surgery; Anesthesia; Pain
Keywords: postoperative pain; general anesthesia; postoperative discomfort
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Nalbuphine; flurbiprofen axetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- flurbiprofen axetil (Active Comparator): flurbiprofen axetil intraoperative administration 100mg
  Interventions: Drug: Flurbiprofen Axetil
- nalbuphine (Experimental): nalbuphine intraoperative administration 0.1mg/kg
  Interventions: Drug: Nalbuphine
- nalbuphine and flurbiprofen axetil (Experimental): flurbiprofen axetil intraoperative administration 100mg and nalbuphine intraoperative administration 0.1mg/kg
  Interventions: Drug: Nalbuphine and Flurbiprofen Axetil

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine administration during surgery
  Arms: nalbuphine
Drug: Flurbiprofen Axetil — Flurbiprofen axetil administration during surgery
  Arms: flurbiprofen axetil
Drug: Nalbuphine and Flurbiprofen Axetil — Nalbuphine and Flurbiprofen Axetil administration during surgery
  Arms: nalbuphine and flurbiprofen axetil

SUMMARY:
The purpose of this study is to evaluate the postoperative pain and discomfort using flurbiprofen axetil or nalbuphine administration after orbital decompression under general anesthesia.

DETAILED DESCRIPTION:
To investigate postoperative analgesia achieved with intraoperative administration of intravenous nalbuphine and flurbiprofen axetil in patients undergoing orbital decompression

ELIGIBILITY:
Inclusion Criteria:

* 16-75 years old
* diagnosed as thyroid eye disease
* bone removal orbital decompression under general anesthesia
* American Society of Anesthesiologists (ASA) physical status of I-II

Exclusion Criteria:

* body mass index (BMI) <18.5 or >35
* any uncontrolled clinical problems

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Pain after orbital decompression | 24 hour after recovery
  Pain levels measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no pain and 10 represents the worst pain imaginable ; this scale has been confirmed to be sensitive and reliable.Clinically significant postoperative pain was considered serious pain (NRS score ≥5).

SECONDARY OUTCOMES:
Discomfort after orbital decompression | 24 hour after recovery
  Discomfort levels were measured using Numerical Rating Scale (NRS) ranging from 0 to 10, where 0 represents no discomfort and 10 represents the worst discomfort; this scale has been confirmed to be sensitive and reliable. Discomfort was defined as "sensation other than pain" and included nausea, vomiting, headache, and dizziness. Clinically significant postoperative discomfort was considered serious discomfort (NRS score ≥5) any time postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Huijing Ye, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided